CLINICAL TRIAL: NCT03908684
Title: Pilot Investigation of Ultrasound Cell Death Imaging and Spectroscopy as Early Indicators of Response to Radiation Treatment in Prostate, Rectum and Head and Neck Cancers, and to Characterize Prostate Masses
Brief Title: Ultrasound Spectroscopy as Early Indicators of Radiation Treatment Response in Prostate, Rectum and Head & Neck Cancers
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Radiation Oncologist and Clinician Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 448-2013
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Head and Neck Cancer; Rectal Cancer
Keywords: Ultrasound; Spectroscopy
MeSH Terms: conditions — Prostatic Neoplasms; Head and Neck Neoplasms; Rectal Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Head and Neck: The research will involve a clinical evaluation consisting of 200 patients in the head and neck cohort. It will assess changes in five different ultrasound spectroscopic parameters over different times during treatment with radiotherapy as predictors of tumour shrinkage and pathologic complete response. Ultrasound parameters investigated will include mid-band fit (related to image intensity), spectroscopic slope (backscatter versus frequency), spectroscopic intercept, histogram fit size and shape parameters which can be used as estimates of scatterer size and concentration.
  Interventions: Device: Ultrasound Imaging
- Prostate: The research will involve a clinical evaluation consisting of 100 patients in the prostate cohort. It will assess changes in five different ultrasound spectroscopic parameters over different times during treatment with radiotherapy as predictors of tumour shrinkage and pathologic complete response. Ultrasound parameters investigated will include mid-band fit (related to image intensity), spectroscopic slope (backscatter versus frequency), spectroscopic intercept, histogram fit size and shape parameters which can be used as estimates of scatterer size and concentration.
  Interventions: Device: Ultrasound Imaging
- Rectum: The research will involve a clinical evaluation consisting of 20 patients in the rectal cohort. It will assess changes in five different ultrasound spectroscopic parameters over different times during treatment with radiotherapy as predictors of tumour shrinkage and pathologic complete response. Ultrasound parameters investigated will include mid-band fit (related to image intensity), spectroscopic slope (backscatter versus frequency), spectroscopic intercept, histogram fit size and shape parameters which can be used as estimates of scatterer size and concentration.
  Interventions: Device: Ultrasound Imaging

INTERVENTIONS:
Device: Ultrasound Imaging — Ultrasound Spectroscopy assess changes in five different ultrasound spectroscopic parameters over different times during treatment with radiotherapy as predictors of tumour shrinkage and pathologic complete response. Ultrasound parameters investigated will include mid-band fit (related to image intensity),spectroscopic slope (backscatter versus frequency), spectroscopic intercept, histogram fit size and shape parameters which can be used as estimates of scatterer size and concentration.
  Other Names: Ultrasound Spectroscopy

SUMMARY:
Our objective in this study is to identify an optimal ultrasound spectroscopy parameter that can be used as an early predictor of pathological complete or partial response in men with prostate cancer and men and women with rectum and head and neck cancers receiving treatment radiotherapy.

We have previously demonstrated that high-frequency ultrasound and spectroscopy, and recently conventional-frequency ultrasound and spectroscopy may be used to detect cell death in vitro, in situ and in vivo. The method can detect different forms of cell death and has been demonstrated to be sensitive to apoptotic, necrotic and mitotic cell death. The main goal, as described above, is to select the best ultrasound spectroscopy parameter to use as an early predictor of pathological complete response

DETAILED DESCRIPTION:
The purpose of the study is to test the hypothesis that ultrasound imaging and spectroscopy may be used as a predictive marker of advanced tumour response to radiotherapy. The main goal is to select the best ultrasound ultrasound spectroscopy parameter and vascular distribution index to use as an early predictor of pathological complete or partial response as a primary endpoint. Tumour size decrease as a secondary endpoint. Other secondary endpoints will include measuring changes in blood vessel distribution with treatment and changes in ultrasound parameters will be correlated with two and five year survival rates. Finally, we will investigate if prostate masses can be characterized (benign vs. malignant) using ultrasound backscatter parameters.

ELIGIBILITY:
Inclusion Criteria:

* (1) Histologically or cytologically confirmed prostate, rectum and head and neck carcinoma which has not been treated with any first-line therapy and will be treated with radiation therapy
* (2) Measurable disease by ultrasound, or MRI performed within 28 days prior to treatment
* (3) Eastern Co-operative Oncology Group (ECOG) Performance Status of 0 or 1
* (4) Life expectancy of at least 6 months
* (5) Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to dosing:

  (i) hemoglobin >90 mg/dL (ii) leukocytes >3,000/mL (iii) absolute neutrophil count >1,500/mL (iv) platelets >100,000/mL (v) total bilirubin within normal institutional limits (vi) AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal (vii) creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional upper limit of normal
* (6) Patients should have the ability to understand and the willingness to sign a written informed consent document. Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* (1) Chemotherapy, radiotherapy, or major surgery within 4 weeks prior to registering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to registration
* (2) Receiving any other investigational agents
* (3) Known brain metastases
* (4) History of allergic reactions attributed to compounds of similar chemical or biologic composition
* (5) Contraindications to radiotherapy such as but not limited to:

  (i) previous radiotherapy to an involved area (ii) active collagen vascular disease (iii) genetic diseases associated with hyper-radiosensitivity
* (6) Any clinically serious infections requiring systemic anti-bacterial, antifungal or antiviral therapy
* (7) Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, and cardiac arrhythmia
* (8) Psychiatric illness/social situations that would limit compliance with study requirements
* (9) History of active ongoing seizure disorder, substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* (10) Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women who are receiving radiotherapy for head and neck cancer, or rectal cancer, and men who are receiving radiotherapy for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2014-12-17 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2029-12-17 (Estimated)

PRIMARY OUTCOMES:
Radiation Treatment Response | Up to 5 years
  Evaluate tumour response to radiotherapy as measured radiologically within the treated therapeutic region.

SECONDARY OUTCOMES:
Radiation Treatment Long-term Clinical Outcome | Up to 5 years
  Evaluating tumour response to radiotherapy as measured radiologically within the treated therapeutic region and assessing long-term clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Osapoetra LO, Dasgupta A, DiCenzo D, Fatima K, Quiaoit K, Saifuddin M, Karam I, Poon I, Husain Z, Tran WT, Sannachi L, Czarnota GJ. Quantitative US Delta Radiomics to Predict Radiation Response in Individuals with Head and Neck Squamous Cell Carcinoma. Radiol Imaging Cancer. 2024 Mar;6(2):e230029. doi: 10.1148/rycan.230029. PMID 38391311
- [Derived] Fatima K, Dasgupta A, DiCenzo D, Kolios C, Quiaoit K, Saifuddin M, Sandhu M, Bhardwaj D, Karam I, Poon I, Husain Z, Sannachi L, Czarnota GJ. Ultrasound delta-radiomics during radiotherapy to predict recurrence in patients with head and neck squamous cell carcinoma. Clin Transl Radiat Oncol. 2021 Mar 12;28:62-70. doi: 10.1016/j.ctro.2021.03.002. eCollection 2021 May. PMID 33778174
- [Derived] Osapoetra LO, Dasgupta A, DiCenzo D, Fatima K, Quiaoit K, Saifuddin M, Karam I, Poon I, Husain Z, Tran WT, Sannachi L, Czarnota GJ. Assessment of clinical radiosensitivity in patients with head-neck squamous cell carcinoma from pre-treatment quantitative ultrasound radiomics. Sci Rep. 2021 Mar 17;11(1):6117. doi: 10.1038/s41598-021-85221-6. PMID 33731738
- [Derived] Dasgupta A, Fatima K, DiCenzo D, Bhardwaj D, Quiaoit K, Saifuddin M, Karam I, Poon I, Husain Z, Tran WT, Sannachi L, Czarnota GJ. Quantitative ultrasound radiomics in predicting recurrence for patients with node-positive head-neck squamous cell carcinoma treated with radical radiotherapy. Cancer Med. 2021 Apr;10(8):2579-2589. doi: 10.1002/cam4.3634. Epub 2020 Dec 13. PMID 33314716